CLINICAL TRIAL: NCT03033693
Title: Study of the Depth of Anesthesia on Postoperative Clinical Outcome in Patients With Supratentorial Tumor
Acronym: DEPTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government); Guiyang Jinyang Hospital (Unknown); Beijing Sanbo Brain Hospital (Other); The Second Hospital of Hebei Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Chinese PLA General Hospital (Other); Anhui Provincial Hospital (Other Government); Guangdong 999 Brain Hospital (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2016-1-20410
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia, Brain Tumor, Supratentorial,Outcome
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The deep anesthesia group (Other)
  Interventions: Other: Bispectral index will be targeted at 35
- The light anesthesia group (Other)
  Interventions: Other: Bispectral index will be targeted at 50

INTERVENTIONS:
Other: Bispectral index will be targeted at 50 — The depth of general anesthesia will be monitored by bispectral index (BIS) at 50.
  Arms: The light anesthesia group
Other: Bispectral index will be targeted at 35 — The depth of general anesthesia will be monitored by bispectral index (BIS) at 35.
  Arms: The deep anesthesia group

SUMMARY:
Recent studies have shown that deep anesthesia is associated with poor outcome. There is still lack of randomized controlled trials with large sample size on the effect of depth of anesthesia on the postoperative outcomes in patients undergoing brain tumor resection. The investigators are performing a randomized and parallel group trial. The aim of the study is to determine whether there is a causal relationship between the depth of anesthesia and postoperative clinical outcome in patients undergoing supratentorial tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive elective supratentorial tumor resection under general anesthesia from 2017 to 2019 will be recruited in the trial. Inclusion criteria include ages between 18 and 80 years old, American Society of Anesthesiologists (ASA) physical status Ⅲ-Ⅳ, surgery duration expected to be equal or more than three hours, postoperative hospital stay expected to be equal or more than five nights, and monitoring BIS throughout anesthesia.

Exclusion Criteria:

* Patients who undergo emergency or awake craniotomy surgery, or unable to present the written consent will be excluded from the trial. The patients whose incision site conflicts with the placement of BIS electrode on the frontal and temporal lobe will also be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1461 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Disability-free survival rate | Postoperative 30 days
  World Health Organization Disability Assessment Schedule 2.0 Scale will be used to assess the body disability. Disability is defined as a 4-point increasement in the WHODAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Study Chair — Department of Anesthesiology, Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Beijing, China

REFERENCES:
- [Derived] Cui Q, Peng Y, Liu X, Jia B, Dong J, Han R. Effect of anesthesia depth on postoperative clinical outcome in patients with supratentorial tumor (DEPTH): study protocol for a randomized controlled trial. BMJ Open. 2017 Sep 11;7(9):e016521. doi: 10.1136/bmjopen-2017-016521. PMID 28899891